CLINICAL TRIAL: NCT01164059
Title: Clinical Effectiveness Of The Newer Antipsychotic Compounds Olanzapine, Quetiapine And Aripiprazole In Comparison With Low Dose Conventional Antipsychotics (Haloperidol And Flupentixol) In Patients With Schizophrenia
Brief Title: Clinical Effectiveness of Newer Antipsychotics in Comparison With Conventional Antipsychotics in Schizophrenia
Acronym: NeSSy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bremen (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Eckart Rüther, Principal Investigator, University of Bremen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NeSSy_200901; 2009-010966-47 (EudraCT Number)
Record Dates: First submitted 2010-07-06; First posted 2010-07-16 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; atypical antipsychotic drugs; conventional antipsychotic drugs; olanzapine; quetiapine; aripiprazole; haloperidol; flupentixol
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; Flupenthixol; Quetiapine Fumarate; Aripiprazole; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atypical antipsychotics (Experimental): Olanzapine, Quetiapine, or Aripiprazole
  Interventions: Drug: Olanzapine; Drug: Quetiapine; Drug: Aripiprazole
- typical antipsychotics (Active Comparator): Haloperidol or Flupentixol
  Interventions: Drug: Flupentixol; Drug: Haloperidol

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 10, 15, or 20 mg / day
  Arms: atypical antipsychotics
Drug: Flupentixol — Flupentixol 6, 9, or 12 mg / day
  Arms: typical antipsychotics
Drug: Quetiapine — Quetiapine 400, 600, or 800 mg / day
  Arms: atypical antipsychotics
Drug: Aripiprazole — Aripiprazole 10, 15, or 20 mg / day
  Arms: atypical antipsychotics
Drug: Haloperidol — Haloperidol 3, 4.5, or 6 mg / day
  Arms: typical antipsychotics

SUMMARY:
This study is designed to compare the efficacy and drug tolerability of two strategies for the treatment of schizophrenia. The two strategies consist of utilizing, on the one hand, a conventional antipsychotic like haloperidol or flupentixol and, on the other hand, a newer antipsychotic compound like olanzapine, quetiapine or aripiprazole in patients with schizophrenia.

DETAILED DESCRIPTION:
There is agreement in the psychiatry community that the so-called atypical antipsychotics should be considered first choice in the treatment of schizophrenic disorders. However, the general superiority of these newer antipsychotic drugs over the older conventional drugs could not be clearly demonstrated in recent controlled clinical trials. The discrepancy between every day's clinical perception and the results of clinical trials raises the question whether the studies performed so far employed the adequate methodological approach to represent the daily practice situation which is characterized by a wide variety of duration and type of the schizophrenic disorder, concomitant diseases, and medications. Moreover, some studies might not have been focused adequately on patient-relevant outcome variables.

The present study project is designed to answer these open questions. The innovative character of the study design is

1. that different neuroleptic strategies will be compared rather than single antipsychotic drugs, using
2. an enhanced biometric design, that provides a choice of treatment with respect to the individual patient though the trial as such is randomised controlled and double blind;
3. that clinically relevant endpoints such as quality of life will be the primary variables, and
4. inclusion and exclusion criteria lead to a study population representing clinical every day practice as near as possible.

Another innovatory procedure is that serum levels of the study drugs will be recorded twice during the study. The authors hope that their design might yield transfer effects for other clinical trials facing similar problems.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* age 18-65 years
* necessity to establish new or change antipsychotic treatment due to unsatisfying results or side effects
* written informed consent

Exclusion Criteria (amongst others):

* Known or suspected hypersensitivity to olanzapine, quetiapine, aripiprazole, flupentixol or haloperidol
* Acute suicidal tendency
* "Einwilligungsvorbehalt (BGB)" or "Unterbringung (PsychKG)"
* Epilepsy
* Organic psychosis
* Parkinson Disease
* Dementia
* History of malignant neuroleptic syndrome
* QTc interval ≥ 0.5s / history of congenital QTc prolongation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2010-02; Primary Completion 2013-08 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Contentment with treatment: Patient (SF-36) | 24 weeks
Contentment with treatment: Psychiatrist (CGI) | 24 weeks

SECONDARY OUTCOMES:
Subscores of SF-36 | 24 weeks
Subjective wellbeing under neuroleptic treatment scale (SWN-K) | 24 weeks
Positive and Negative Syndrome Scale (PANSS) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- Germany (18):
  - Universitätsklinikum Aachen, Aachen
  - Krankenhaus Angermünde, Angermünde
  - Karl-Jaspers-Klinik, Bad Zwischenahn
  - Charité - Universitätsmedizin Berlin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - LWL-Universitätsklinik Bochum der Ruhr-Universität, Bochum
  - Klinikum Bremen-Ost gGmbH, Bremen
  - Rheinische Kliniken Düsseldorf der Heinrich-Heine-Universität, Düsseldorf
  - Städtisches Krankenhaus Eisenhüttenstadt GmbH, Eisenhüttenstadt
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Privat-Nerven-Klinik Dr. med. Kurt Fontheim, Liebenburg
  - Dietrich-Bonhoeffer-Klinik Neubrandenburg, Neubrandenburg
  - Ruppiner Kliniken, Neuruppin
  - Ernst von Bergmann Klinikum, Potsdam
  - Immanuel Klinik Rüdersdorf, Rüdersdorf
  - Klinik Taufkirchen, Taufkirchen

REFERENCES:
- [Derived] Ibragimov K, Keane GP, Carreno Glaria C, Cheng J, Llosa AE. Haloperidol (oral) versus olanzapine (oral) for people with schizophrenia and schizophrenia-spectrum disorders. Cochrane Database Syst Rev. 2024 Jul 3;7(7):CD013425. doi: 10.1002/14651858.CD013425.pub2. PMID 38958149
- [Derived] Veselinovic T, Scharpenberg M, Heinze M, Cordes J, Muhlbauer B, Juckel G, Habel U, Ruther E, Timm J, Grunder G; NeSSy Study Group. Disparate effects of first and second generation antipsychotics on cognition in schizophrenia - Findings from the randomized NeSSy trial. Eur Neuropsychopharmacol. 2019 Jun;29(6):720-739. doi: 10.1016/j.euroneuro.2019.03.014. Epub 2019 Apr 10. PMID 30981585
- [Derived] Grunder G, Heinze M, Cordes J, Muhlbauer B, Juckel G, Schulz C, Ruther E, Timm J; NeSSy Study Group. Effects of first-generation antipsychotics versus second-generation antipsychotics on quality of life in schizophrenia: a double-blind, randomised study. Lancet Psychiatry. 2016 Aug;3(8):717-729. doi: 10.1016/S2215-0366(16)00085-7. Epub 2016 Jun 2. PMID 27265548
- [Derived] Schulz C, Timm J, Cordes J, Grunder G, Muhlbauer B, Ruther E, Heinze M. Patient-oriented randomisation: A new trial design applied in the Neuroleptic Strategy Study. Clin Trials. 2016 Jun;13(3):251-9. doi: 10.1177/1740774516639910. Epub 2016 Mar 25. PMID 27016729